CLINICAL TRIAL: NCT06197165
Title: Amylo-Shiatsu-Acute-Chronic: Effects of Shiatsu on Symptoms and Quality of Life of Amyloidosis Patients
Acronym: AMYLO-SHIATSU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP230424
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Amyloidosis
Keywords: Cardiac amyloidosis - Targeted Shiatsu - pain
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shiatsu (Experimental): Comfort Shiatsu: 39
  Targeted Shiatsu: 39
  Interventions: Other: Targeted Shiatsu
- without Shiatsu (Active Comparator): patients with cardiac amyloidosis with severe symptoms
  Interventions: Other: Targeted Shiatsu

INTERVENTIONS:
Other: Targeted Shiatsu — demonstrate the beneficial impact targeted Shiatsu compared with a "comfort" Shiatsu

SUMMARY:
The objective of this study is to assess the beneficial effects of three targeted Shiatsu sessions compared to "comfort" Shiatsu on symptoms in patients with severe cardiac amyloidosis. Specifically, the study aims to evaluate the short-term impact of a targeted Shiatsu session on neuro-cardiovascular physiological parameters and symptoms in patients with cardiac amyloidosis, in comparison to comfort Shiatsu and no Shiatsu. Additionally, the study will investigate the effects of three targeted Shiatsu sessions versus "comfort" Shiatsu and no Shiatsu on various symptoms (fatigue, sleep disturbances, pain, anxiety, depression, dyspnea, digestive disorders, nausea) and quality of life in cardiac amyloidosis patients with severe symptoms. Patient satisfaction with Shiatsu will also be evaluated, alongside an assessment of the tolerance to Shiatsu.

DETAILED DESCRIPTION:
IAmyloidosis leads to a wide range of disorders, including vascular, cardiac, neuropathic, digestive, renal, and others. These impairments significantly affect patients' quality of life, autonomy, and are often accompanied by stress and anxiety. Literature reviews indicate that complementary approaches have a positive impact on alleviating the symptoms of disabling chronic illnesses, with Shiatsu showing efficacy in several international studies. As part of an initiative to improve patient care and better address their chronic, persistent symptoms, we propose incorporating Shiatsu targeted specifically at amyloidosis symptoms as a complementary therapy. How can Shiatsu help patients with amyloidosis? What impact does it have on their quality of life and various symptoms?

Hypothesis/Objective:

This study aims to demonstrate the beneficial impact of three targeted Shiatsu sessions compared to "comfort" Shiatsu on symptoms in cardiac amyloidosis patients with severe symptoms. Additionally, it will assess the short-term effects of a targeted Shiatsu session on neuro-cardiovascular physiological parameters and symptoms in cardiac amyloidosis patients, comparing the effects of targeted Shiatsu, comfort Shiatsu, and no Shiatsu. The study will evaluate the impact of these interventions on symptoms such as fatigue, sleep disturbances, pain, anxiety, depression, dyspnea, digestive disorders, and nausea, as well as the overall quality of life. It will also assess patient satisfaction with Shiatsu and evaluate the therapy's tolerance.

Method:

This is a randomized, controlled, superiority, single-center, double-blind study comparing the effects of "targeted" Shiatsu sessions on amyloidosis symptoms with those of "comfort" (non-targeted) Shiatsu sessions.

Population:

The study will involve patients diagnosed with amyloidosis (TTR, WT, AL) who are hospitalized or followed at the Centre de Référence Amyloses-Cardiaques (Cardiogen branch) at the CHU Henri Mondor in Créteil, France. A total of 108 patients will participate: 78 in the Shiatsu group (26 AL, 26 TTR, 26 WT), 39 in the Comfort Shiatsu group, 39 in the Targeted Shiatsu group, and 30 in the No Shiatsu group. The expected inclusion rate per center per month is 4.5, with a study duration of 2 years.

Primary Endpoint:

Reduction in total ESAS symptom score 48 hours after the third Shiatsu session.

Secondary Endpoints:

A 20% improvement in heart rate variability measured with the e-patch. A 20% improvement in skin conductance and variability measured with the SUDOSCAN.

Overall score on the EQ-5D scale. Overall score on the MINNESOTA scale. A 2-point improvement in the symptom-specific questionnaire corresponding to the symptom targeted by Shiatsu (e.g., dyspnea, digestive disorders, pain).

Improvement in at least one global score on the BFI, HADS, or LSEQ scales.

Inclusion Visit (D0):

Patients will be offered participation during their routine care consultation. Once consent is obtained, the patient will complete several questionnaires (MINNESOTA, EESE-R, EQ-5D, QCD, BFI, LSEQ, HADS). Measurements with the SUDOSCAN will be taken, and the e-patch will be applied for 48 hours. For Shiatsu participants, randomization will be conducted by an open-label CRA independent of the study, and the results will be sent to the Shiatsu specialists (targeted or comfort). The patient will then receive a Shiatsu session accordingly.

Research Follow-Up Visits:

Visit 1 (D1): A second SUDOSCAN measurement will be taken 24 hours post-Shiatsu session or inclusion for the no-Shiatsu group. Follow-up measurements will be taken at 24 and 48 hours.

Visit 2 (D2): A third SUDOSCAN measurement will be taken 48 hours post-Shiatsu or inclusion. Patients will complete the EESE-R and modified TAQ questionnaires.

Visit 3 (D7±1 day): The Shiatsu group will receive a second Shiatsu session and complete the modified TAQ questionnaire 48 hours later (D9±1 day).

Visit 4 (D14±1 day): The Shiatsu group will receive a third Shiatsu session and complete the modified TAQ questionnaire 48 hours after the session (D16±1 day).

Telephone Visits:

Contact 1 (D16±1 day): Telephone follow-up 48 hours after the third Shiatsu session, during which patients will complete various questionnaires (MINNESOTA, EESE-R, EQ-5D, QCD, BFI, LSEQ, HADS, modified TAQ).

Contact 2 (D31±1 day): A second telephone follow-up to complete the same set of questionnaires.

Conclusion:

The expected benefits for patients include an improvement in quality of life and symptoms (e.g., appetite, nausea, digestive disorders, sleep, fatigue, anxiety, depression, pain) as well as balancing of the autonomic nervous system (ANS), which is often weakened by disease progression and hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years ;
* Patient with :

  * Transthyretin of genetic origin (TTR) ;
  * Transthyretin of non-mutated origin (WT) ;
  * Light Chain (AL);
* Membership of a social security scheme, beneficiary or beneficiary's beneficiary (excluding AME);
* Written patient consent.
* Score greater than or equal to 3 on the EESE-R questionnaire (Edmonton Symptom Evaluation Scale-Revised), for at least 1 symptom among: dyspnea, digestive disorders, nausea, pain, anxiety, depression (Shiatsu and non-Shiatsu groups);
* Score global à l'EESE-R supérieur ou égal à 10 (groupes Shiatsu et sans shiatsu).

Exclusion Criteria:

* Patients with orthostatic hypotension;
* Patients with bullous amyloidosis (fragile skin);
* Patients who have already received Shiatsu treatment;
* Patient with insufficient autonomy to maintain sitting position;
* Patient with insufficient autonomy to move from home to hospital;
* Participating in another interventional study, or within the exclusion period of a previous study, if applicable;
* Known pregnancy or breast-feeding;
* Patient under known guardianship at the time of inclusion;
* Patient under AME.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-04-12 (Estimated); Study Completion 2026-04-12 (Estimated)

PRIMARY OUTCOMES:
EESE-R (ESAS) TOTAL SYMPTOM SCORE AT 48 HOURS AFTER THIRD SHIATSU SESSION | 31 days ± 1 day
  Description of efficacy endpoints for primary endpoint: Reduction in total ESAS symptom score at 48 hours after third shiatsu session. Questionnaire at J0 (before first session) - J2 (48 H after first session)- J16 48H (after third session) - J31 48H (15 days after third session).

SECONDARY OUTCOMES:
MEASUREMENT PHYSIO, SUDOSCAN, E-PATCH | 48 hours
  Description of secondary endpoint: 20% improvement in heart rate variability measured with the e-patch. Continuous measurement [0-48H] after first Shiatsu session

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU HENRI MONDOR, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION